CLINICAL TRIAL: NCT01919463
Title: Intubation Techniques on Colonoscopy Quality: A Single Center Randomized Control Clinical Trial
Brief Title: Intubation Techniques on Colonoscopy Quality (SINOCOLO2013)
Acronym: SINOCOLO2013
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, En-Da Yu, Surgical Professor, Vice Director of Department of Colorectal Surgery and Center of GI Endoscopy, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SINOCOLO2013
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Adenoma; Colorectal Polyp
Keywords: Colonoscopy; Lower Gastrointestinal Tract; Magnetic Endoscopic Imaging; Abdominal Compression
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): Colonoscopy is completed without abdominal compression by GI assistants. Live image of magnetic endoscopic imaging system is shown to investigators for study but not to the colonoscopist for facilitating the intubation process.
- Experimental Group 2 (Monitoring) (Experimental): Colonoscopy is completed with abdominal compression by GI assistants. Live image of magnetic endoscopic imaging system is shown to investigators for study but not to the colonoscopist for facilitating the intubation process. The colonoscopist directs GI assistants to conduct compression by his subjective judgement.
  Interventions: Behavioral: Abdominal Compression
- Experimental Group 1 (Guiding) (Experimental): Colonoscopy is completed with abdominal compression by GI assistants. Live image of magnetic endoscopic imaging system is shown both to investigators for study and to the colonoscopist for facilitating the intubation process. The colonoscopist directs GI assistants to conduct compression according to the guidance of magnetic endoscopic imaging system.
  Interventions: Behavioral: Abdominal Compression; Device: Guidance of Magnetic Endoscopic Imaging (MEI) System

INTERVENTIONS:
Behavioral: Abdominal Compression — Abdominal Compression is conducted by GI assistants during intubation process to facilitate the process. It can be conducted at different ares of the abdomen with different force.
  Arms: Experimental Group 1 (Guiding); Experimental Group 2 (Monitoring)
Device: Guidance of Magnetic Endoscopic Imaging (MEI) System — Live image of MEI can show the form of the colonoscope inside the body. Live image is show to colonoscopist for facilitating the intubation process.
  Other Names: MEI System (Olympas, Tokyo, Japan)
  Arms: Experimental Group 1 (Guiding)

SUMMARY:
The primary aim of this study is

- to explore the usefulness of abdominal compression on intubation.

Other aims include

1. to investigate the effectiveness and the efficacy of different manners of abdominal compression and to analysis the reasons of their success and failure
2. to get the knowledge of the formation of colon loops and its frequency
3. to clarify the impact of intubation with loops on adenoma detection rate

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo colonoscopy examination for screening, surveillance, diagnosis or treatment

Exclusion Criteria:

* Pregnant female patients
* Patients who have history of colorectal cancer, colorectal polyposis, inflammatory bowel disease or heredity colorectal neoplasm syndrome such as familiar adenomatous polyposis, Lynch Syndrome and so on
* Patients who had previous abdominal surgery
* Patients who are known to have colonic stricture or obstructing tumor from the results of radiography (X ray, CT scan or barium enema)
* Patients who are presenting acute surgical conditions such as severe colitis, megacolon and active gastrointestinal bleeding
* Patients who have inadequate bowel preparation
* Patients who reject to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-08 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Mean Intubation Time (MIT) | At the end of the procedure, up to 1 hour
  MIT refers to the mean of intubation time. Intubation time refers to the time spent on the intubation procedure. Intubation is defined as the procedure during which the tip of the colonoscope reaches the cecum from the anus.

SECONDARY OUTCOMES:
Cecal Intubation Rate (CIR) | At the end of the procedure, up to 1 hour
  CIR refers to the proportion of the subjects who receive the whole colon examination. The whole colon examination means the tip of the colonoscope reaches the cecum during the procedure.
Pain Score (PS) | During the procedure, up to 1 hour
  PS is measure by the numerical rating scale during the intubation process. Numerical rating scale contains 11 ranks from 0 to 10, in which 0 means no pain and 10 means the extreme pain cannot be borne.
Severe Adverse Event Rate (SAER) | The day of the procedure, 24 hours
  SAER refers to the proportion of the subjects to whom severe adverse events happens. Severe adverse events include perforation, massive hemorrhage, lethal arrhythmia, death and so on.
Adenoma Detection Rate (ADR) | At the end of the procedure, up to 1 hour
  ADR refer to the rate of adenoma detection, calculated as the proportion of subjects with at least one adenoma.
Polyp Detection Rate (PDR) | At the end of the procedure, up to 1 hour
  PDR refer to the rate of polyp detection, calculated as the proportion of subjects with at least one polyp.

CONTACTS AND LOCATIONS:
Overall Officials: En-Da Yu, M.D., Principal Investigator — Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Shah SG, Saunders BP, Brooker JC, Williams CB. Magnetic imaging of colonoscopy: an audit of looping, accuracy and ancillary maneuvers. Gastrointest Endosc. 2000 Jul;52(1):1-8. doi: 10.1067/mge.2000.107296. PMID 10882954
- [Background] Holme O, Hoie O, Matre J, Stallemo A, Garborg K, Hasund A, Wiig H, Hoff G, Bretthauer M. Magnetic endoscopic imaging versus standard colonoscopy in a routine colonoscopy setting: a randomized, controlled trial. Gastrointest Endosc. 2011 Jun;73(6):1215-22. doi: 10.1016/j.gie.2011.01.054. Epub 2011 Apr 8. PMID 21481862
- [Background] Cheung HY, Chung CC, Kwok SY, Tsang WW, Li MK. Improvement in colonoscopy performance with adjunctive magnetic endoscope imaging: a randomized controlled trial. Endoscopy. 2006 Mar;38(3):214-7. doi: 10.1055/s-2005-921172. PMID 16528645